CLINICAL TRIAL: NCT03183531
Title: New Protocol for Identification of Serious Bacterial Infection in Febrile Newborn
Brief Title: New Protocol for Febrile Neonate Management
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Bulbul, Associate professor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: sislietfal.06.2017
Record Dates: First submitted 2017-06-06; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Newborn; Infection; Newborn Sepsis
MeSH Terms: conditions — Infections; Neonatal Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: C reactive protein — Addition of C-reactive protein test for management strategies to follow-up febrile neonates in outpatient.

SUMMARY:
The objective of present study was to evaluate clinical and laboratory characteristics of febrile neonate and describe the incidence of SBI in febrile neonates. Secondarly investigators aimed to test usefulness of major protocols and new protocol in evaluating only febrile neonate.

DETAILED DESCRIPTION:
This was a prospective observational cohort study, conducted between January 2011 and December 2015 (5 years) at Sisli Hamidiye Etfal Hospital, a tertiary care university-affiliated medical center in Istanbul. Written informed consent was obtained from the parents of all infants enrolled in the study before inclusion. The study protocol was approved by the local ethic committee.

Study population All neonates who were admitted to the neonatal intensive care unit with a rectal temperature of ≥38°C (documented at the time of medical evaluation) were eligible for the participation in this study. The exclusion criteria were gestational age less than 35 weeks, who refused to participate in the study, chromosome abnormality (e.g., trisomy 21, 18), the presence of a chronic disease, congenital malformations (cyanotic heart disease, meningomyelocele), admission to pediatric surgery, started on antibiotics before admission, and incomplete records. A complete history was obtained from the parents of infants, and a specialist in neonatology carried out a physical examination for localizing the source of the fever in all infants.

Data collection The data obtained for all infants included: demographic information (age at admission, gender, and birth weight), general assessment (well or sick-appearing), medical history, physical examination findings, laboratory test results, and final diagnosis. Laboratory investigations including complete blood count, CRP level, blood chemistry and culture, urine sample analysis and culture (obtained by bladder catheterization), and cerebrospinal fluid sample analysis and culture, were carried out. In the presence of respiratory symptoms or signs, chest radiography was performed. Lumbar puncture was performed according to the ward's policy, which is required for every infant if neurologic findings are positive or without the focus on fever. Stool specimens were obtained when a history of diarrhea was noted and sent for white blood cell analysis and bacterial culture. Other tests were conducted as necessary. Skin, soft tissue, and ear infections were diagnosed by physical examination.

Definition of SBI An episode of SBI was defined as (A) the growth of a known pathogenic bacteria in one or more of cultures (bacteremia, meningitis, osteomyelitis, suppurative arthritis, urinary tract infection, bacterial enteritis, and pneumonia), (B) any disease commonly associated with bacterial pathogens including pneumonia, acute otitis media, suppurative arthritis, osteomyelitis, and soft-tissue infections (cellulitis, abscess, mastitis, and omphalitis). Pneumonia was defined as a new discrete infiltration on the chest film, which was confirmed by an attending pediatric radiologist with the presence of typical clinical signs and symptoms.

All specimens for culture were evaluated by standard microbiological methods. No specimens were processed for viral cultures. The blood culture isolates were considered pathogenic if the organism was known to cause disease in healthy infants. UTI (urinary tract infection) was defined as the isolation of >104 CFU/mL of urine of a single pathogen by catheterization. A positive urine analysis was defined by a positive test for leucocyte esterase or nitrite by the dipstick method or leukocyte ≥10 cells/mm3 in uncentrifuged urine. Methods of viral agent evaluation: in infants with viral respiratory symptoms and complaints (a runny nose, sneezing, coughing), the presence of RSV-Ag (rapid immunochromatographic test produced by Prima lab SA, Switzerland), and influenza-Ag (Immunoassay test produced by Dalian Rongbang Medical Healthy Devices, Spain) were assessed from nasopharyngeal secretions. The body weight of the subjects was taken on admission and weight loss was assessed according to the birth weight. The proportion of weight loss more than twelve percent of birth weight was considered as dehydration.

All patients were hospitalized and prophylactic antibiotic therapy was started and continued for at least 72 hours (cases diagnosed only with dehydration did not receive antibiotics).

Newly proposed protocol (Sisli Etfal) includes:

(1) Unremarkable medical history (no perinatal antibiotics, no underlying disease, not hospitalized longer than the mother), (2) Good appearance, (3) No focal physical signs of infection, (4) CRP level < 1 mg/dl, (5) WBC 5000-15000 counts/mm3 and band/neutrophil ratio (I/T) <0.2, (6) A normal urine analysis.

The infants with all these criteria were considered to have a low risk for SBI. All infants were classified at low-risk by the criteria of Rochester, Boston, Philadelphia and Sisli Etfal protocols. The criteria of four protocols are presented in Table 1.

Statistical analysis The data were analyzed by using SPSS version 15.0 (SPSS, Chicago, IL, USA). Categorical variables are reported as percentages, and normally distributed data are expressed as mean±SD. Statistical comparisons between two groups performed with Student's t-test for normally distributed data, Mann-Whitney U test for non-normally distributed data, and chi-square test for all numerical and categorical values. The positive predictive value (PPV) for SBI of at least one abnormal criteria and the NPV for SBI of the low-risk criteria, in combination, were calculated by the standard statistical formula. All patients were evaluated according to the Boston, Philadelphia, Rochester and Sisli Etfal protocols, and the results were compared for sensitivity, specificity, NPV, PPV, and accuracy values. For predicting SBI, the serum levels of CRP and WBC count were subjected to receiver operating characteristics (ROC) curve analysis. The results were considered to be significant if analysis yielded p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* All neonates who were admitted to the neonatal intensive care unit with a rectal temperature of ≥38°C (documented at the time of medical evaluation) were eligible for the participation in this study.

Exclusion Criteria:

* The exclusion criteria were gestational age less than 35 weeks, who refused to participate in the study, chromosome abnormality (e.g., trisomy 21, 18), the presence of a chronic disease, congenital malformations (cyanotic heart disease, meningomyelocele), admission to pediatric surgery, started on antibiotics before admission, and incomplete records.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborn babies admitted to hospital with fever
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of characteristics of febrile neonate and describe the incidence of SBI in febrile neonates. | 5 years
  All febrile neonate admitted and evaluated for SBI. An episode of SBI was defined as (A) the growth of a known pathogenic bacteria in one or more of cultures (bacteremia, meningitis, osteomyelitis, suppurative arthritis, urinary tract infection, bacterial enteritis, and pneumonia), (B) any disease commonly associated with bacterial pathogens including pneumonia, acute otitis media, suppurative arthritis, osteomyelitis, and soft-tissue infections (cellulitis, abscess, mastitis, and omphalitis). Pneumonia was defined as a new discrete infiltration on the chest film, which was confirmed by an attending pediatric radiologist with the presence of typical clinical signs and symptoms.
Usefulness of major protocols and new protocol in evaluating only febrile neonate. | 5 years
  All infants were classified at low-risk by the criteria of Rochester, Boston, Philadelphia and new created Sisli Etfal protocols.

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Etfal Education and Research Hospital, Istanbul, Turkey (Türkiye)